CLINICAL TRIAL: NCT05348512
Title: Laborstudie Zur Aufnahme Spektraler Und Photoplethysmographischer Daten
Brief Title: Laboratory Study for the Acquisition of Spectral and Photoplethysmographic Data
Acronym: LabStud_MSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Ines Gockel, Univ.-Prof. Dr. med., MBA, University of Leipzig
Other Study IDs: LabStud_MSI/iPPG
Record Dates: First submitted 2022-04-07; First posted 2022-04-27 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: spectral imaging — non-contact, non-invasive hyperspectral and multispectral imaging without a diagnostic test
Other: photoplethysmography — non-invasive pulse oximetry without a diagnostic test

SUMMARY:
Laboratory study on healthy volunteers to acquire spectral video data from the tongue and fingers as well as photoplethysmographic data from the forehead, fingers, and earlobes to evaluate and optimize algorithms for imaging photoplethysmography (iPPG) and multispectral imaging (MSI)

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers >= 18 years old

Exclusion Criteria:

* pregnant and nursing women
* persons unable to consent
* persons with tattoos or diseases on the tongue, finger, ear, or forehead
* narcoleptics
* epileptics
* persons with arterial hypertension, peripheral arterial disease, anemia, Raynaud syndrome, autoimmune vasculitides, Takayasu arteritis, venous insuffiencies, microangiopathy, diabetic vasculopathy, scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers >= 18 years
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
RGB video data | 16 minutes
  true color video data (10 bit per channel [red, green, blue]) from tongues and fingers
hyperspectral data | 16 minutes
  false color parameter images, representing the oxygenation in %; the perfusion; the hemoglobin, water, and fat content of tissue in arbitrary units betwenn 0 and 100 from tongues and fingers (imaged areas have to correspond to RGB video data)
multispectral video data | 16 minutes
  true color video data (10 bit per channel [red, green, blue]) from tongues and fingers (imaged areas have to correspond to RGB video data)
plethysmographic wave | 5 minutes
  numerical value in arbitrary values representing the amount of transmitted/reflected light over time through fingers or earlobes or from the forehead
pulse | 5 minutes
  frequency in bpm (beats per minute) or Hz (Hertz)
pulsation index | 5 minutes
  ratio between pulsating and non-pulsating tissue components in %
SpO2 | 5 minutes
  oxygenation of arterial blood in %, measured with a pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Ines Gockel, Prof. Dr., Principal Investigator — University of Leipzig
Locations (1):
- Department of Visceral, Transplantation, Vascular and Thoracic Surgery, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared. However, results are planned to be published in a scientific journal in a completely anonymized manner.